CLINICAL TRIAL: NCT02796274
Title: Historical Case Record Survey of Visual Acuity Data From Patients With Leber's Hereditary Optic Neuropathy (LHON)
Status: Completed | Type: Observational
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SNT-CRS-002
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Leber's Hereditary Optic Neuropathy (LHON)
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The purpose of this survey is to collect visual acuity data from patients with LHON in order to establish the clinical course (natural history) and visual acuity outcomes in patients with a genetically confirmed diagnosis of LHON. In addition, this survey will generate data that will serve as comparator for the open-label study SNT-IV-006.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 12 years
2. the onset of symptoms is dated after 1999 and is well documented (at least month of onset of symptoms is known for each eye)
3. at least two VA assessments are available within 5 years of onset of symptoms and prior to idebenone use
4. have a genetic diagnosis for LHON for one of the following mitochondrial DNA (mtDNA) mutations: G11778A, G3460A, T14484C

Exclusion Criteria:

1. any participation in an interventional clinical trial after the onset of symptoms
2. any other cause of visual impairment (e.g. glaucoma, diabetic retinopathy, AIDS related visual impairment, cataract, macular degeneration, etc.) or any active ocular disorder (uveitis, infections, inflammatory retinal disease, thyroid eye disease, etc.) during the data collection period

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a genetically confirmed diagnosis of LHON
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2016-05; Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klopstock, Prof. Dr., Principal Investigator — Friedrich-Baur-Institut, Muenchen, Germany
Locations (21):
- Belgium (4):
  - CHU Saint-Pierre, Brussels
  - Cliniques Universitaire Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - C. H. U. Sart Tilman, Liège
- France (5):
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - Hopital Roger Salengro - CHU Lille, Lille
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - CHU Reims - Hôpital Robert Debré, Reims
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg
- Germany (3):
  - Justus-Liebig-Universitaet Giessen, Giessen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Friedrich-Baur-Institut, München
- Italy (4):
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Università di Pisa, Pisa
  - G. B. Bietti Fondazione - IRCCS, Rome
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Oogziekenhuis Rotterdam, Rotterdam
- Haukeland Universitetssykehus, Bergen, Norway
- United Kingdom (2):
  - University Hospital of Wales, Cardiff
  - Queen's Hospital, London

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- LHON Patients Case Record Cohort: Historical case record data from all LHON patients fulfilling the prospectively-defined inclusion criteria:
  1. Age ≥ 12 years.
  2. Onset of symptoms was dated after 1999 and was well documented (at least month of onset of symptoms is known for each eye).
  3. At least two VA assessments were available within 5 years of onset of symptoms and prior to idebenone use.
  4. Have a genetic diagnosis for LHON for one of the following mtDNA mutations: G11778A, G3460A, or T14484C.
Period: Overall Study
Arm/Group | LHON Patients Case Record Cohort
Started | 219; 438 eyes
Completed | 219; 438 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Visual Acuity (VA) at Baseline (logMAR)
Units Other Than Participants: eyes
Groups:
- LHON Patients Case Record Cohort: Historical case record data from all LHON patients fulfilling the prospectively-defined inclusion criteria:
  1. Age ≥ 12 years.
  2. Onset of symptoms was dated after 1999 and was well documented (at least month of onset of symptoms is known for each eye).
  3. At least two VA assessments were available within 5 years of onset of symptoms and prior to idebenone use.
  4. Have a genetic diagnosis for LHON for one of the following mtDNA mutations: G11778A, G3460A, or T14484C.
  Actual: 48 (with VA assessment made ≤1 year after the onset of symptoms) out of 219 patients from whom data were collected and entered into the database.
Arm/Group | LHON Patients Case Record Cohort
Number analyzed (Participants) | 219
Number analyzed (eyes) | 438
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49
  Between 18 and 65 years | 169
  >=65 years | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26.0 [18.0 to 41.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 175
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 24
  Belgium | 30
  Poland | 40
  Italy | 20
  United Kingdom | 20
  France | 29
  Germany | 56

OUTCOME MEASURES:

1. Primary Outcome: In Eyes With VA Assessment Made ≤1 Year After Onset of Symptoms: Proportion of Eyes With Clinically Relevant Recovery (CRR) of VA (Measured by Change in ETDRS Letters) From Baseline (BL) or in Which BL VA Better Than 1.0 logMAR Was Maintained at 12 Months
Description: Clinically Relevant Recovery (CRR) is defined as a VA improvement from off-chart (ETDRS) to 5 letters on-chart, or an on-chart improvement of 10 letters.
Time Frame: 12 months
Population: Data from a total of 219 LHON patients and 438 eyes were obtained from this study, out of which 96 eyes had a VA assessment made ≤1 year after the onset of symptoms (primary outcome measure).
Measure: Median (Inter-Quartile Range); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | LHON Patients Case Record Cohort
Number analyzed (Participants) | 219
Number analyzed (eyes) | 96
ETDRS letters | 15 [1.5 to 34.5]

ADVERSE EVENTS:
Time Frame: No safety data was collected
Description: No safety data was collected
Arm/Group | LHON Patients Case Record Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT02796274/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT02796274/SAP_001.pdf